CLINICAL TRIAL: NCT05013411
Title: Rethinking Observations in Mental Health
Status: Completed | Type: Observational
Sponsor: Oxehealth Limited (Industry)
Collaborators: Central and North West London NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 295362
Record Dates: First submitted 2021-08-12; First posted 2021-08-19 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Vital Signs
Keywords: Nurse Observations; Clinical Observations

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthcare workers: Healthcare workers with patient care experience and are willing to share their experience of current practices of obtaining patient observations.
  Interventions: Other: Qualitative study

INTERVENTIONS:
Other: Qualitative study — Individual interviews and focus groups will be conducted to explore current strengthens and barriers in obtaining patient observations. Views on use of technology in assisting with patient observations will also be discussed and documented.

SUMMARY:
To gain healthcare workers' perception of the current observations practices used in patient care and explore the benefits of using technology to enhance observations in inpatient mental health setting in the United Kingdom.

DETAILED DESCRIPTION:
Periodic intermittent clinical observations are commonly used in mental health services at admission for risk assessment and then for the clinical management of patients.

Nurses follow these practices as routine care to ensure patient well-being. However, being observed may make patients feel uncomfortable and anxious.

The Department of Health (2006) stipulated for the practice of observation to be implemented in a manner that would enable patients to experience it as a healing and compassionate practice. This is apparently not always realised as there are reported differences on how patients are observed, and clinical data obtained.

Whilst this may be attributed in part to lack of or limited training on the use of observations, it can also in part be attributed to lack of a standardised approach to implementation and documentation of the outcomes of observations (Stewart & Bowers 2012).This contributes to variability among healthcare workers in their interpretation of the outcomes/data of observations. Given that patients' care pathways are influenced by the outcomes/data of observations, it is critical to reduce the variability in the use of this practice. Doing so would lead to obtaining consistent and dependable data that reflect patients' mental state to guide their individual care pathways.

The focus of this qualitative study is to document how clinicians perform routine patient observations, the essential aspects of observations through a clinician's point of view and how can application of modern technology aid this process. This systematic documentation will capture the strengths and limitations of current practice creating a service provide based dataset to inform focused improvements.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers such as nurse directors, matrons, ward managers, nurses, healthcare support workers, including; nurse associates, nurse assistants and assistant practioners who work in inpatient mental health settings
* Healthcare workers with at least two years' experience of working in inpatient mental settings
* Healthcare workers who conduct or have conducted patient observations, and have used it for at least two years

Exclusion Criteria:

Students and clinicians in training who do not carry out independent patient observations.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Healthcare workers with experience of taking patient observations in inpatient mental health setting in the UK
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Strengthens and Limitations of current practice of clinical observations | Day 1 of participation, during a one-off interview/focus group
  Exploratory method, conducted in the form of individual and focus groups to document strengthens and barriers to current ways of obtaining clinical observations in in patient mental health setting.(qualitative method)

SECONDARY OUTCOMES:
Views on use of technology in obtaining patient observations | Day 1 of participation, during a one-off interview/focus group
  Exploratory method to gain healthcare workers' perspective on using modern technology such as a contact free patient monitoring system to aid the practice of patient observations through individual interviews and focus groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ade Odunlade, Principal Investigator — Central North West London NHS Foundation Trust
Locations (1):
- Ade Odunlade, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Quotes maybe shared making reference to participant's job descriptions.